CLINICAL TRIAL: NCT05845918
Title: PRogram to Improve Stress-levels and Enhance Memory
Acronym: PRISEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ambar Kulshreshtha, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004811; 1K23AG066931-01A1 (NIH); 2025P011143 (Other: Emory IRB)
Record Dates: First submitted 2023-03-27; First posted 2023-05-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment
Keywords: lifestyle intervention; Chronic Stress
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRISEM Remote (Experimental): PRISEM Remote is a remote-based lifestyle intervention program in which participants will attend 17 core online sessions via Zoom from the evidence-based Diabetes Prevention Program curriculum with remaining post-core sessions to reinforce strategies and activities introduced in the core program for the duration of 6 months.
  Interventions: Behavioral: PRISEM Remote

INTERVENTIONS:
Behavioral: PRISEM Remote — Participants will attend 1-hour sessions weekly for 12 weeks (12 sessions) then biweekly for 8 weeks (4 sessions) and 1 session in the last month (1 session). Sessions will be group-based and will cover the following topics: 1) Program Overview, 2) Get Active, 3)Track Activity, 4) Eating Well, 5) Track Food, 6) Get More Active, 7) Energy In, Energy Out, 8) Eating to Support Health Goals, 9) Manage Stress, 10) Eat Well Away From Home, 11) Managing Triggers, 12) How to Stay Active, 13) Take Charge of Thoughts, 14) Get Back on Track, 15) Get Support (from friends and family), and 16) Staying Motivated. Sessions will include a brief presentation of the topic, followed by an introduction to tools and strategies to practice. This is a facilitated program with participants "driving" the direction and acting as peer support to one another.

SUMMARY:
This is a pilot study with the objective to examine if an in-person and a remote multi-component intervention program can improve chronic stress, vascular measures, and executive function among African American and White patients with Mild Cognitive Impairment. Researchers plan to enroll 45 participants with over-recruitment of African American patients. Participants will be recruited to participate in PRogram to Improve Stress-levels and Enhance Memory (PRISEM) (i.e., remote lifestyle intervention program). The participants will be asked to participate in group-based and/or individual activities that focus on improving health education, nutrition, physical activity, cognitive health, stress levels, and overall well-being. The duration of the study for all participants will be 12 months with 3 study visits. At each study visit, the following measures will be assessed: psychosocial, behavioral, vascular/physical, and executive function.

DETAILED DESCRIPTION:
More than half the patients with Mild Cognitive Impairment (MCI), a transitional state between normal aging and dementia, will develop dementia within five years. Despite the clinical and public health significance of MCI, there are no known pharmacological treatment strategies preventing the progression to Alzheimer's Disease (AD). Disappointing results from clinical trials of AD-modifying interventions have increased efforts to focus on prevention strategies that delay the onset of the disease. Since AD-related pathology begins more than a decade before patients develop symptoms, prevention efforts are likely to be more effective when targeted earlier in life. Data is even more limited on higher-risk groups, such as African Americans, who have double the incidence compared with Whites.

This study plans to enroll a diverse population with an over-enrollment of African Americans because African Americans have a higher risk of developing mild cognitive impairment (MCI) and double the incidence of Alzheimer's Disease (AD) compared with Whites. Unfortunately, the prevention and management of MCI have been understudied among African Americans. Chronic stress (such as perceived discrimination and daily environmental stress) in African Americans can affect cognition and plays a role in the worsening of unhealthy behaviors such as smoking, improper diet, and physical inactivity.

Recent studies have predicted that a 10-25% reduction in seven key modifiable risk factors, including behavioral and lifestyle choices, could prevent 1.3 million AD cases globally. Healthy lifestyle approaches can reduce oxidative stress, produce structural and functional changes in the brain, and also influence the rate of neurogenesis in adult and senescent animal models. However, interventions that improve these have often been disappointing, in part because the impact of each lifestyle behavior on AD risk is relatively small.

This pilot study aims to evaluate how a remote multicomponent lifestyle intervention program improves mood symptoms (chronic stress) and positively impacts biomarkers of vascular health and the autonomic nervous system among forty African American and White patients with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 years or older
* Fluency in English
* African American or White
* MCI will be defined as subjective memory complaints with a Montreal Cognitive Assessment (MoCA) 19- 25
* Prior diagnosis of MCI
* Participants would be sedentary at baseline (self-report of <30 minutes of structured physical activity <3 times per week in the last 6 months) and have poor Mediterranean-Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet scores (using the MIND diet screener)

Exclusion Criteria:

* Dementia diagnosis or reversible causes of dementia (e.g., if the patient has hypothyroidism or low vitamin B12 that is contributing to the subject's cognitive impairment)
* Active medical or psychiatric diseases that in the judgment of the investigator would affect the safety of the subject or scientific integrity of the study (e.g., actively manic patient)
* Uncontrolled medical conditions, such as congestive heart failure, reflected by poor exercise tolerance and shortness of breath
* Any physical ailment, such as stroke with residual impairment, that is a barrier to performing study procedures and attending sessions
* History of brain lesions, stroke, or major head trauma in the past year
* Those who are unable to demonstrate that they understood the details of the study (i.e., lack of decisional- capacity to consent) or linguistic limitations
* Pregnant women, prisoners, and adults unable to consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility for the PRISEM pilot to collect additional stress and vascular measurements | 6 months
  Feasibility will be calculated as the percentage of participants who agree to participate and are enrolled according to the target, with a loss to follow-up.
Acceptability for the PRISEM pilot to collect additional stress and vascular measures. | Baseline, 6 months, and 12 months
  Acceptability of the PRISEM pilot participants will be assessed using semi-structured interviews regarding vascular and stress measures conducted over the course of the study.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) score | Baseline, 6 months, and 12 months
  The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all 10 scale items. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Short Form (SF)-12 Quality of Life (QoL) score | Baseline, 6 months, and 12 months
  The SF-12 QoL uses two items each to estimate scores for four to eight health concepts (physical functioning, role-physical, role-emotional, and mental health). Scores for the remaining four health concepts (bodily, pain, general health, vitality, and social functioning) are estimated using one item each. The lower the score the more disability.
Weight | Baseline and 6 months
  Self-reported weight (Kg) will be collected at each study time point
Body Mass Index (BMI) | Baseline and 6 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI will be calculated at each study time point.
Systolic and diastolic blood pressure (BP) measurements | Baseline and 6 months
  Systolic and diastolic blood pressure (SBP and DBP)will be measured at each time point. BP (mmHg) will be assessed by utilizing an automatic sphygmomanometer in which a cuff will be placed on the participant's forearm.
Heart rate variability (HRV). | Baseline and 6 months
  Heart rate variability (HRV) will be measured with an ECG monitor. A validated signal processing code will be used to evaluate these signals for noise and detect the necessary ECG component measures, and when outliers are suspected, a visual inspection will be performed. If any episodes of Atrial fibrillation are detected by the program, they will be confirmed by the study team and excluded. HRV will be examined in 5-minute sliding windows, and the median, 10th percentile, and minimum values will be calculated.
Pulse Wave Analysis. | Baseline and 6 months
  Indices of arterial stiffness and wave reflections will be estimated in the supine position using the Sphygmocor device (Atcor Medical, Australia), which records sequential high-quality pressure waveforms at peripheral pulse sites using a high-fidelity tonometer. Pulse-wave velocity (PWV) measured between carotid and femoral arteries is a regional assessment of aortic stiffness and is the gold standard index of arterial stiffness.
Trail Making Test (TMT) Part A | Baseline, 6 months, and 12 months
  The TMT is a measure of attention, speed, and mental flexibility. It also tests spatial organization, visual pursuits, recall, and recognition. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part A tests visual scanning, numeric sequencing, and visuomotor speed. A score over 78 seconds may indicate a deficit in visual perception. The average time is around 29 seconds.
Trail Making Test (TMT) Part B | Baseline, 6 months, and 12 months
  Trail Making Test (TMT) Part B is scored based on the time in seconds it takes to complete the task, which involves alternating between connecting numbered and lettered circles in ascending order (1-A-2-B-3-C). Part B assesses cognitive flexibility and executive function, and is scored separately from Part A. A higher score indicates greater cognitive impairment.
Flanker Test | Baseline, 6 months, and 12 months
  The Flanker test measures inhibitory control and attention by having participants identify a central stimulus (fish or arrows) while ignoring flanking stimuli. Scoring is based on both accuracy and reaction time. If a participant's accuracy is below 80% correct, the score is based solely on accuracy. If accuracy is 80% or higher, both accuracy and reaction time are used to calculate the score. This ensures participants who are accurate but slow, or fast but inaccurate, are scored accordingly. The final computed score is converted to an age-adjusted scale score. A score of 100 represents the national average for a given age, with 115 being one standard deviation above average and 85 being one standard deviation below average.
Pattern Comparison Processing Speed Test (PCPST) | Baseline, 6 months, and 12 months
  PCPST is an assessment of processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same. It measures how quickly a person can decide if two visual patterns are identical, scoring how many correct comparisons are made in a set time. Scores are converted to normative scores that compare performance to a representative sample, with a higher score indicating better processing speed. A mean of 100 with a standard deviation of 15 is considered average, with scores indicating the test-taker's performance relative to their age group or the general population.
Picture Sequence Memory (PSM) test | Baseline, 6 months, and 12 months
  The Picture Sequence Memory (PSM) test, specifically the NIH Toolbox version, is scored by counting the number of adjacent pairs of pictures correctly placed in the sequence across three learning trials. The meaning of the score is that it provides a measure of episodic memory, which is the ability to recall and place in order a series of events or images. A higher score indicates better episodic memory performance, while lower scores suggest memory impairments.
List Sorting Working Memory Test scores | Baseline, 6 months, and 12 months
  The List Sorting Working Memory Test scores are calculated based on the number of stimuli correctly recalled and sequenced in order of size. The test has two phases: a one-dimensional phase (1-List) and a two-dimensional phase (2-List). A higher score indicates better working memory, meaning an individual can better register, maintain, and manipulate visual and auditory information.
Dimensional Change Card Sort (DCCS) | Baseline, 6 months, and 12 months
  The Dimensional Change Card Sort (DCCS) measures cognitive flexibility by assessing how well a person can switch between different sorting rules. It typically involves sorting cards by one rule (e.g., color) and then switching to a new rule (e.g., shape). The test records how many cards are correctly sorted and how long it takes to respond. Pass/Fail: The primary scoring method is a pass/fail based on performance after the rule-switching "switch" trials.
Physical Activity Scale for the Elderly (PASE) | Baseline and 6 months
  The PASE score (Physical Activity Scale for the Elderly) is a numerical value derived from a 12-item questionnaire that measures the physical activity level of older adults over the past week. Meaning is determined by the score, with higher scores indicating greater physical activity. Scores are calculated by multiplying the frequency, duration, and intensity of various activities (leisure, household, occupational) by pre-determined weights and summing them up, resulting in a score that can range from 0 to 400 or more.
  Interpreting scores: Sedentary: 0-40; Light Physical Activity: 41-90; Moderate to Intense Activity: 91+
Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet Quiz | Baseline, 6 months, and 12 months
  The MIND diet quiz is a 15-point assessment of how closely participants' diet aligns with the MIND (Mediterranean-DASH Intervention for Neurodegenerative Delay) eating plan. The final score, which ranges from 0 to 15, indicates their level of adherence and is associated with their potential for better cognitive health. Higher scores (above 9): Indicate they are following the MIND diet closely.
  Moderate scores (7 and 8): Suggest a moderate alignment with the MIND diet. Even moderate adherence has been shown to provide a reduced risk of Alzheimer's compared to the lowest scores.
  Lower scores (below 6): Indicate that their diet is less aligned with the brain-healthy principles of the MIND diet.

CONTACTS AND LOCATIONS:
Overall Officials: Ambar Kulshreshtha, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Goizueta Alzheimer's Disease Research Center (GADRC), Atlanta, Georgia
  - Emory Dunwoody Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share deidentified individual participant data that underlie published articles.
Supporting Information: Study Protocol
Time Frame: The investigators will share deidentified individual participants beginning 9 months and ending 2 years following article publication
Access Criteria: The investigators will share deidentified individual participant data with researchers who provide a methodologically sound proposal to achieve the aims of the approved proposal.
  Please direct inquiries to mindandheart@emory.edu

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT05845918/ICF_000.pdf